CLINICAL TRIAL: NCT03599895
Title: Combined Application of 3D Printing Technology and Robotic Surgery in Radical Gastrectomy of Gastric Cancer
Brief Title: Application of 3D Printing Technique in Radical Gastrectomy With Leonardo da Vinci Robot
Acronym: 3DINGCRS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XJTU1AF-3D-2017-006
Record Dates: First submitted 2018-07-17; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Stomach Neoplasms
Keywords: 3D printing technology
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D printing group (Experimental): the radical gastrectomy for gastric cancer of Davinci robotic surgery with the assistance of 3D printing model
  Interventions: Procedure: 3D printing model
- non 3D printing group (Experimental): the radical gastrectomy for gastric cancer of Davinci robotic surgery without the assistance of 3D printing model
  Interventions: Procedure: non 3D printing model

INTERVENTIONS:
Procedure: 3D printing model — Combine the 3D printing technique with imaging examination ,making the 3D model of da Vinci robot assisted radical gastrectomy
  Arms: 3D printing group
Procedure: non 3D printing model — da Vinci robot assisted radical gastrectomy
  Arms: non 3D printing group

SUMMARY:
The incidence of gastric cancer is the highest in China, and surgery is one of the most effective treatment methods. Da Vinci robot radical gastrectomy for gastric cancer has the advantage of minimally invasive and fine operation. However, due to complicated perigastric anatomy, abundant blood supply and wide distribution of lymph nodes, it is widely used in clinical use of .Combine the 3D printing technique with imaging examination (digestive endoscopy,3Dct cta/ctv, etc.) ,making the 3D model of da Vinci robot assisted radical gastrectomy can fully show the anatomical relationship around gastric cancer, determine the flow and variation of splenic portal vessels, and the distribution of splenic hilar lymph nodes. In order to eliminate the imagination difference of spatial anatomical structure before operation, it is easier for surgeons to optimize the operation plan, to control the operation process and to improve the accuracy, and to adopt individualized operation suitable for the patients.

DETAILED DESCRIPTION:
The investigators will work with general surgery, imaging department and 3D printing center to try to print gastric cancer model and guide the operation. After obtaining the approval of the Hospital Ethics Committee, 20 patients with gastric cancer were collected for imaging examination and evaluation, and the normal physical model of 70% normal volume was printed with Guang Min resin material.The investigators will analyse the anatomical relationship between the tumor and surrounding tissues,and determine the range of tumor excision and the feasibility and safety of radical gastrectomy with Leonardo da Vinci robot for gastric cancer.Through the assistance of the 3D model,The investigators will select the suitable operation path to determine the extent of tumor excision and lymph node dissection.Furthermore, 3D print model is used to provide real-time navigation for key steps of surgery. The purpose of this research is to observe the application value of 3D printing technique in gastric cancer laparoscopic surgery with Leonardo da Vinci robot radical gastrectomy, and to provide reference for the development of 3D printing model of other complicated digestive tract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients without contraindications gastroscope，surgery and anesthesia;
* There is no history of abdominal surgery, no severe abdominal cavity adhesion;
* Not found the tumor metastasis;
* Normal coagulation function;
* There is no history of anticoagulant drugs, or who take aspirin, salvia miltiorrhiza, etc., should stop taking drugs for more than one week;
* Patients and their families volunteered choice the surgical procedure and signed informed consent.

Exclusion Criteria:

* Patients with preoperative assessment of distant metastasis;
* Patients with preoperative radiation and chemotherapy or hormone therapy;
* Patients with acute obstruction, bleeding or perforation of the emergency surgery;
* Patients with a history of abdominal trauma or abdominal surgery;
* Patients with contraindications gastroscope，surgery and anesthesia.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-03-30 (Estimated)

PRIMARY OUTCOMES:
operation time | 1 hours to 6 hours through the surgery completion
  record in minutes,from the beginning of anesthesia to the end

SECONDARY OUTCOMES:
blood loss | 1 hours to 6 hours through the surgery completion
  from the surgical record sheet
success rate | from two days to two weeks after surgery
  the time in bed to the postoperative patient
time in bed | from two days to two weeks after surgery
  the time in bed to the postoperative patient
time to take food | from two days to two weeks after surgery
  the time to eat to the postoperative patient
postoperative complication rate | from two weeks to one year after surgery
  including anastomotic stoma fistula,anastomotic stenosis,abdominal
tumor recurrence rate | from one month to 2 years after surgery
  periodic review the CT or MRI or endoscope
hospitalization expenses | 1 month
  total hospitalization expenses